CLINICAL TRIAL: NCT04691141
Title: A Phase I/II, Open-label Study to Investigate the Pharmacokinetics, Safety, and Efficacyof ATG 016 Monotherapy in IPSS-R Intermediate Risk and Above Myelodysplastic Syndrome (MDS) Patients After Failure of Hypomethylating Agent (HMA)-Based Therapy
Brief Title: A Study to Evaluating the Pharmacokinetics, Safety, and Efficacy of ATG 016 Monotherapy in IPSS-R Intermediate Risk and Above Myelodysplastic Syndrome (MDS)
Acronym: HATCH
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped early because the sponsor decided to change the study-drug development strategy
Sponsor: Shanghai Antengene Corporation Limited (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-016-MDS-001
Record Dates: First submitted 2020-12-23; First posted 2020-12-31 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-016 (Experimental): 5 mg QD×Days 1-5/week will be the initial dose of this study.
  Interventions: Drug: ATG-016

INTERVENTIONS:
Drug: ATG-016 — 59 patients enrolled will be treated with ATG-016, orally, each 4 week (28-day) a cycle

SUMMARY:
This is a Phase Ⅰ/II, Open-label Study to Investigate the Pharmacokinetics, Safety, and Efficacyof ATG 016 Monotherapy in IPSS-R Intermediate Risk and above Myelodysplastic Syndrome (MDS) Patients after Failure of Hypomethylating Agent (HMA)-based Therapy.

DETAILED DESCRIPTION:
This is a Phase Ⅰ/II, Open-label Study to Investigate the Pharmacokinetics, Safety, and Efficacyof ATG 016 Monotherapy in IPSS-R Intermediate Risk and above Myelodysplastic Syndrome (MDS) Patients after Failure of Hypomethylating Agent (HMA)-based Therapy. In Phase I: approximately 15 to 21 subjects and Phase II: approximately 44 subjects; approximately 59 to 65 subjects will be enrolled totally in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
2. ≥18 years of age, males or females.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
4. A life expectancy longer than 3 months in the opinion of the investigator at the screening.
5. Male subjects (Including those who have received vasectomy) must agree to use condoms during sex with a woman of childbearing age and have no plans to impregnate the woman throughout the study and for 3 months following the last dose after the date of signing the ICF.

Exclusion Criteria:

1. History of central nervous system (CNS) involvement.
2. Toxicity from prior antitumor therapy did not return to Grade 1 or baseline (Except for alopecia, neutropenia, anemia, and thrombocytopenia. For neutrophils, hemoglobin, and platelets, please follow Exclusion Criteria No. 5).
3. History of human immunodeficiency virus (HIV) infection.
4. History of severe bleeding disorder, such as hemophilia A, hemophilia B, and vascular hemophilia.
5. History of allogeneic stem-cell transplantation.
6. Serious psychiatric or medical conditions that, in the opinion of the investigator, could interfere with treatment, compliance, or the ability to give consent.
7. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
MTD in Phase I | 16 months
  MTD will be evaluated using the NCI-CTCAE, Version 5.0
RP2D in Phase I | 16 months
  RP2D will be determined under the guidance of the SRC.
AEs/SAEs | 25 months
  Toxicity will be graded according to the NCI CTCAE, Version 5.0.
ORR in Phase II | 25 months
  Based on 2006 IWG Response Criteria, evaluated by IRC: ORR (CR + PR + mCR)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) in Phase I/II | 12 months
  DCR (CR + PR + mCR + HI + SD)
Duration of Response (DOR) in Phase I/II | 12 months
  To evaluate duration of response
Progression-Free Survival (PFS) in Phase I/II | 12 months
  To evaluate progression-free survival
Overall Survival (OS) | 12 months
  The estimates of Kaplan-Meier

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Xiao, MD, Principal Investigator — Tianjin blood research institute
Locations (6):
- China (6):
  - Guangdong Provincal People's Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai the sixth people's hospital, Shanghai, Shanghai Municipality
  - Tianjin blood research institute, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang